CLINICAL TRIAL: NCT04652570
Title: A Phase 1b/2a Study of VB119 in Adult Subjects With Primary Membranous Nephropathy
Brief Title: Efficacy and Safety of VB119 in Subjects With Membranous Nephropathy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor change
Sponsor: Tenet Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 119-01-01
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VB119 dose escalation (Experimental): Dose escalation phase followed by a dose expansion phase. VB119 to be administered as intravenous infusions.
  Interventions: Drug: VB119

INTERVENTIONS:
Drug: VB119 — Humanized, immunoglobin (Ig) G1 monoclonal antibody (mAb) to be administered as intravenous infusion at multiple timepoints during the study.

SUMMARY:
This study is a Phase 1b/2a, open-label, sequential-cohort, dose escalation, and dose expansion study to evaluate the safety, tolerability, PK, and PD of VB119 in subjects with primary MN

ELIGIBILITY:
Inclusion Criteria:

1. Is ≥ 18 years of age at the time of informed consent;
2. Has a kidney biopsy-proven diagnosis of primary MN within the past 10 years; Note: It is preferable that subjects enrolled have kidney biopsy tissue samples that are positive for anti-PLA2R antibody staining. Subjects with kidney biopsy-proven diagnosis of primary MN >10 years and ≤20 years that meet all other eligibility criteria may be enrolled after discussion with the Medical Monitor.
3. 3. Has a documented laboratory history of nephrotic range proteinuria (defined as either greater than or equal to 3.5 g total protein per 24-hour urine collection or greater than or equal to 3.5 g/g UPCR by spot collection) AND has proteinuria with a UPCR greater than or equal to 2.0 g/g based on 2 consecutive spot urine (first morning void) sample collections obtained within 14 days of each other during the Screening Period. Both samples must qualify;
4. Has systolic blood pressure (BP) <160 mmHg or diastolic BP <100 mmHg after 5 minutes of rest at Screening;
5. Is willing and able to provide written informed consent prior to Screening;
6. Female subjects of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone in the postmenopausal range at Screening, based on the central laboratory's ranges;
7. Female subjects of childbearing potential (ie, ovulating, premenopausal, or not surgically sterile) and all male subjects must use a medically accepted, highly effective contraceptive regimen during their participation in the study and for 125 days after the last administration of study drug.
8. Male subjects must agree to abstain from sperm donation through 125 days after administration of the last dose of study drug.

Exclusion Criteria:

1. Has an eGFR <45 mL/min/1.73 m2 at Screening utilizing the Chronic Kidney Disease Epidemiology Collaboration formula confirmed by the central laboratory;
2. Has an absolute neutrophil count <1.5 x 10/L;
3. Has a white blood cell count <3.0 x 10/L;
4. Has secondary causes of MN (eg, malignancy, hepatitis B or C, human immunodeficiency virus [HIV], systemic lupus erythematosus [SLE], or other autoimmune diseases [eg, thyroiditis], drug-induced);
5. Has a diagnosis or history of SLE (including non renal disease);
6. Has type 1 or 2 diabetes mellitus;
7. Has an acute, chronic, or latent infection, including tuberculosis, hepatitis, HIV, or chronic urinary tract infections;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 18 months
  Safety and Tolerability
Incidence of Clinical Laboratory Assessments | Through study completion, an average of 18 months
  Safety and Tolerability

SECONDARY OUTCOMES:
% of Patients with Anti-Drug Antibodies | Through study completion, an average of 18 months
Maximum Plasma Concentration [Cmax] | Week 12
Time to Maximum Plasma Concentration [Tmax] | Week 12
% of patients achieving complete remission of proteinuria | Through study completion, an average of 18 months
Anti-PLA2R Antibody Assessment | Through study completion, an average of 18 months
Quality of Life as assessed by PROMIS | Through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Keenan, Study Chair — ValenzaBio, Inc.
Locations (4):
- United States (4):
  - Clinical Reserach Site, Los Angeles, California
  - Clinical Research Site, Albany, New York
  - Clinical Research Site, Bethlehem, Pennsylvania
  - Clinical Research Site, Dallas, Texas